CLINICAL TRIAL: NCT02593045
Title: Open Label, Multicenter Phase I Study of IPH4102, a Humanized Anti-KIR3DL2 Monoclonal Antibody, in Patients With Relapsed/Refractory Cutaneous T-cell Lymphomas (CTCL)
Brief Title: Study of IPH4102 in Patients With Relapsed/Refractory Cutaneous T-cell Lymphomas (CTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH4102-101
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2019-02

CONDITIONS: Cutaneous T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPH4102 (Experimental)
  Interventions: Biological: IPH4102

INTERVENTIONS:
Biological: IPH4102

SUMMARY:
The primary objective of this first in human study is to assess the safety and tolerability of increasing intravenous (IV) doses of single agent IPH4102 administered to patients with relapsed/refractory CTCL to characterize the dose limiting toxicities (DLT) and identify a Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed/refractory, biopsy-proven primary cutaneous T-cell lymphoma who have received at least two previous standard systemic therapies and, if MF/SS, is stage IB IVB at study entry.
2. Centrally assessed KIR3DL2 expression on tumor cells.
3. Patients must have the following minimum wash-out from previous treatments:

   * ≥12 weeks for total skin electron beam irradiation,
   * ≥4 weeks for monoclonal antibodies (≥8 weeks for alemtuzumab),
   * ≥3 weeks for local radiation therapy, systemic cytotoxic anticancer therapy, treatment with other anti-neoplastic investigational agents
   * ≥3 weeks for systemic retinoids, interferons, vorinostat, romidepsin, fusion proteins
   * ≥3 weeks for phototherapy
   * ≥2 weeks for topical therapy (including steroids, retinoids, nitrogen mustard or imiquimod) Topical steroids (maximum strength: medium potency) and oral steroids (≤10 mg prednisone equivalent/day) are allowed, if the patient has been on a stable dose with stable symptoms for at least 4 weeks prior to study entry.
4. At least 18 years of age.
5. ECOG performance status of ≤2.
6. Adequate baseline laboratory data: hemoglobin >9 g/dL, absolute neutrophil count (ANC) ≥1,000/µL, CD4+ T-cells ≥200/µL, platelets ≥50,000/µL, bilirubin ≤1.5 X upper limit of normal (ULN) or ≤3 X ULN for patients with Gilbert's disease, serum creatinine ≤1.5 X ULN, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3 X ULN.
7. Women of childbearing potential (WOCBP) must have a negative serum beta-HCG pregnancy test result within seven days of treatment and must practice an effective method of contraception during treatment and for at least 9 months (270 days) following the last dose of study drug.
8. Female patients who are post-menopausal or surgically sterile.
9. Male patients who agree to practice effective barrier contraception.
10. Ability to understand and the willingness to sign a written informed consent document.
11. No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

1. Patients with limited disease (if MF/SS: stages IA) or central nervous system (CNS) disease.
2. Clinical relevant AEs or laboratory results related to previous anti-neoplastic therapy have not resolved to a NCI-CTCAE grade ≤1.
3. Concomitant corticosteroid use, systemic or topical, for treatment of skin disease. However, topical steroids (maximum strength: medium potency) and oral steroids (≤10 mg prednisone equivalent/day) are allowed, if patient has been on a stable dose with stable symptoms for at least 4 weeks prior to study entry.
4. Patients who have undergone major surgery <4 weeks prior to starting study drug.
5. Patients who have undergone a stem cell transplantation.
6. Patients with known NCI CTCAE Grade 3 or higher (requiring IV antibiotics) active systemic or cutaneous viral, bacterial, or fungal infection.
7. Patients who are Hepatitis B or Hepatitis C antibody positive.
8. Patients who are known to be HIV-positive.
9. Prior hypersensitivity reaction to monoclonal antibodies, other therapeutic proteins, or immunotherapy.
10. Patients with a history of other malignancies during the past three years. (The following are exempt from the three-year limit: non-melanoma skin cancer, Lymphomatoid papulosis, curatively treated localized prostate cancer, curatively treated localized breast cancer, resected thyroid cancer, biopsy proven cervical intraepithelial neoplasia or cervical carcinoma in situ).
11. Patients who are currently pregnant or breastfeeding.
12. Patients with congestive heart failure, Class III or IV, by New York Heart Association (NYHA) criteria.
13. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment.
14. Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLT) | Within 2 weeks after the first administration

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Stanford Cancer Center, Stanford, California
  - Ohio State University, Columbus, Ohio
- Hôpital Saint-Louis, Paris, France
- Leiden University Medical Center, Leiden, Netherlands
- Guy's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Bagot M, Porcu P, Marie-Cardine A, Battistella M, William BM, Vermeer M, Whittaker S, Rotolo F, Ram-Wolff C, Khodadoust MS, Bensussan A, Paturel C, Bonnafous C, Sicard H, Azim HA Jr, Kim YH. IPH4102, a first-in-class anti-KIR3DL2 monoclonal antibody, in patients with relapsed or refractory cutaneous T-cell lymphoma: an international, first-in-human, open-label, phase 1 trial. Lancet Oncol. 2019 Aug;20(8):1160-1170. doi: 10.1016/S1470-2045(19)30320-1. Epub 2019 Jun 25. PMID 31253572